CLINICAL TRIAL: NCT03725085
Title: An Open Label, Multicentric Study to Evaluate the Safety and Tolerability of Mucinex™(Guaifenesin) 600 mg Extended-Release Bi- Layer Tablets in the Treatment of Otherwise Healthy Patients With Symptoms of Cough, Thickened Mucus and Chest Congestion
Brief Title: Study to Evaluate the Safety and Tolerability of Mucinex™(Guaifenesin) 600 mg Extended-Release Bi-Layer Tablets in the Treatment of Otherwise Healthy Patients With Symptoms of Cough, Thickened Mucus and Chest Congestion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Reckitt Benckiser LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-MUC-PMS-IN
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-02

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mucinex™ (GGE, 600 mg extended-release bi-layer tablets) (Experimental): 2 tablets of Mucinex™ (GGE, 600 mg ER bi-layer tablets, taken as 1200 mg BID dose) every 12 hours (twice daily, in the morning and the evening) orally with a full glass of water for 7 days.
  GGE = Guaifenesin
  BID = Twice in a day
  Interventions: Drug: Mucinex™ extended-release (SE)

INTERVENTIONS:
Drug: Mucinex™ extended-release (SE) — 2 tablets of Mucinex™ (GGE, 600 mg extended-release bi-layer tablets)
  Other Names: Guaifenesin bi-layer tablet

SUMMARY:
This was an open label, multicentric, non-comparative, single arm prospective post marketing surveillance (PMS) study to evaluate the safety and tolerability of Mucinex™ (GGE, 600 mg ER bi-layer tablets, taken as 1200 mg BID dose) in the treatment of otherwise healthy patients with symptoms of cough, thickened mucus and chest congestion due to URTI. Symptomatic patients who visited the outpatient department of hospitals and clinics or general physicians and had agreed to participate in this study were screened and enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

Patients were eligible for enrolment in the study if they fulfilled the following criteria:

1. Males and females (non-pregnant) patients of ≥ 18 years of age.
2. Otherwise healthy patients suffering from cough with symptoms of thickened mucus and chest congestion and a diagnosis of any one of the following:

   * Acute Bronchitis
   * Upper Respiratory Tract Infections (URTI) such as naso-pharyngitis
   * Sinusitis
3. Females of child bearing potential:

   1. Must have used efficacious and reliable method of contraception during the entire duration of the study {e.g. double barrier methods (e.g., condom and spermicidal); intrauterine device (IUD) } or remained sexually inactive throughout the study*.
   2. Must have had a negative urine pregnancy test (UPT) at Screening/Baseline (test must have a sensitivity of at least 25 mIU/mL for HCG).
   3. Must have been non-lactating.
4. Patients must have demonstrated their willingness to participate in the study and comply with the study procedures and required visits.
5. Patients must have been willing to authorize use and disclosure of protected health information collected for the study.
6. Patients must have had the ability to understand and sign a written consent, which had to be signed prior to study specific procedures being performed.

   * *Abstinence (sexually inactive) was not an acceptable form of contraception; however, abstinent female patients could have been admitted to the study if they agreed, and signed a statement to the effect, that upon becoming sexually active, they would use a condom with spermicide from that time through 30 days beyond completion of the study (Visit 2).

Exclusion Criteria:

Patients were excluded from the study if they fulfilled any of the following:

1. Females who were pregnant or lactating or planning to become pregnant during the study period.
2. Patients with a history of chronic cough of > 3 weeks duration.
3. Patients with any of the following conditions:

   * Asthma
   * Chronic bronchitis
   * Emphysema
   * Other chronic pulmonary conditions such as Chronic Obstructive Pulmonary Disease (COPD) or cystic fibrosis (CF), etc.
4. Patients with known hypersensitivity to GGE.
5. Patients with temperature greater than 101°F (38.3°C) at Screening/Baseline.
6. Patients with a serious and/or uncontrolled medical condition (chronic or active liver disease, renal impairment, heart disease, diabetes, severe respiratory disease, rheumatoid arthritis, current malignancies, immunocompromised conditions or any other disease) that in the opinion of the investigator would interfere with the study or place the patient at unacceptable risk.
7. Patients with a history or examination findings of alcohol dependence, alcohol or drug abuse or suspected abuse within the past 2 years.
8. Patients who had participated in a study of an investigational drug within 30 days prior to the Screening/Baseline visit.
9. Patients who in the opinion of the investigator were unable to comply fully with the study requirements.
10. Related to persons involved directly or indirectly with the conduct of this study [i.e., investigator, sub-investigators, study coordinators, other study personnel, employees of Reckitt Benckiser or Ecron AcuNova Ltd. (EAL), formerly known as Manipal Acunova Limited (MAL) and the families of each].

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2015-01-24 (Actual); Primary Completion 2015-10-16 (Actual); Study Completion 2015-10-16 (Actual)

REFERENCES:
- [Derived] Tripathi S, Nikhare A, Sharma G, Shea T, Albrecht H. Safety And Tolerability Of Extended-Release Guaifenesin In Patients With Cough, Thickened Mucus And Chest Congestion Associated With Upper Respiratory Tract Infection. Drug Healthc Patient Saf. 2019 Oct 10;11:87-94. doi: 10.2147/DHPS.S222109. eCollection 2019. PMID 31632154

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a multicentric study conducted in 9 study centres across 7 cities in India.
Pre-assignment Details: A total of 554 subjects were screened, 552 subjects enrolled and 550 of them completed the study.
Groups:
- Mucinex™: Subjects received a twice daily dose of Mucinex™ 600 mg Guaifenesin extended-release bi-layer tablets every 12hours
Period: Overall Study
Arm/Group | Mucinex™
Started | 552
Completed | 550
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Mucinex™
Number analyzed (Participants) | 552
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.3 (15.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203
  Male | 349
Height [Mean (Standard Deviation); unit: cms] | 160.8 (8.25)
Weight [Mean (Standard Deviation); unit: Kgs] | 62.5 (11.08)
Race [Count of Participants; unit: Participants]
  Asian | 552
  others | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events (AEs), Type of AE(s) and Frequency of AE(s)
Description: Treatment Emergent Adverse Event (TEAE) are events occurring after the first dose of study medication.
  Frequency of AE(s) - the total Number of Events
  Type of AE(s) - Serious TEAE and Non serious TEAE
Time Frame: Up to Day 9
Population: Safety Population: All patients enrolled in the study were included for safety analyses.
Measure: Number; unit: Number of Events
Arm/Group | Mucinex™
Number analyzed (Participants) | 552
Number of Events
  Treatment Emergent Adverse Event (TEAE) | 29
  Serious TEAE | 0
  Non serious TEAE | 29
  Number of Events | 29

2. Primary Outcome: Number of Subjects Affected With Adverse Events
Description: Proportion of patients with AE(s) - Number of Subjects affected with Events
Time Frame: Up to Day 9
Population: Safety Population: All patients enrolled in the study were included for safety analyses.
Measure: Number; unit: Number of Subjects affected with Events
Arm/Group | Mucinex™
Number analyzed (Participants) | 552
Number of Subjects affected with Events | 28

3. Primary Outcome: Number of Adverse Events by Severity, Seriousness and the Relationship of AE(s) to Treatment
Description: Intensity determined. Mild = AE did not limit usual activities; subject may have experienced slight discomfort.
  Moderate = AE resulted in some limitation of usual activities; subject may have experienced significant discomfort.
  Severe = AE resulted in an inability to carry out usual activities; subject may have experienced intolerable discomfort/pain.
  Relationship to Investigational Medicinal Products (IMP) Unassessable/Unclassified = Insufficient information to be able to make an assessment Conditional/ Unclassified = Insufficient information to make an assessment at present Unrelated = No possibility that the AE was caused by the IMP Unlikely = Slight, but remote, chance that the AE was caused by the IMP, but the balance of judgment was that it was most likely not due to the IMP.
  Possible = Reasonable suspicion that the AE was caused by the IMP Probable = Most likely that the AE was caused by the IMP Certain = AE was definitely caused by the IMP
Time Frame: Up to Day 9
Population: Safety Population: All patients enrolled in the study were included for safety analyses.
Measure: Number; unit: Number of Events
Arm/Group | Mucinex™
Number analyzed (Participants) | 552
Number of Events
  Treatment Emergent Adverse Event (TEAE) | 29
  Serious TEAE | 0
  TEAE Leading to Withdrawal | 0
  TEAE by severity: Mild | 29
  TEAE by severity: Moderate | 0
  TEAE by severity: Severe | 0
  Relationship to IMP - Certain | 0
  Relationship to IMP - Probable | 5
  Relationship to IMP - Possible | 13
  Relationship to IMP - Unlikely | 3
  Relationship to IMP - Unrelated | 8
  Relationship to IMP - Conditional/Unclassified | 0
  Relationship to IMP - Unassessable/Unclassifiable | 0

4. Secondary Outcome: Overall Assessment of the Study Medication by End of Study Patient Questionnaire
Description: End of Study Patient Questionnaire is a questionnaire provided to the patients for overall assessment of the study medication at the end of study visit.
  Satisfied(stfd) Dissatisfied(Dstfd)
Time Frame: Up to Day 9
Population: Safety Population: All patients enrolled in the study were included for safety analyses.
Measure: Count of Participants; unit: Participants
Groups:
- Mucinex™: Subjects received a twice daily dose of Mucinex™ 600mg Guaifenesin extended-release bi-layer tablets every 12hours
Arm/Group | Mucinex™
Number analyzed (Participants) | 552
Participants
  Improvement of Chest Congestion: Very Satisfied | 95
  Improvement of Chest Congestion: Satisfied | 379
  Improvement of Chest Congestion: Mostly Satisfied | 67
  Improvement of Chest Congestion: Not Satisfied | 9
  Improvement of Chest Congestion: Missing | 2
  Improvement of Chesty Cough: Very Satisfied | 97
  Improvement of Chesty Cough: Satisfied | 372
  Improvement of Chesty Cough: Mostly Satisfied | 73
  Improvement of Chesty Cough: Not Satisfied | 8
  Improvement of Chesty Cough: Missing | 2
  First Improvement: During 1st Day of Treatment | 75
  First Improvement: At 2 Days Of Treatment | 360
  First Improvement: Within 3 Days of Treatment | 95
  First Improvement: More than 3 Days of Treatment | 20
  First Improvement: Missing | 2
  Dosing easy to take / convenient: Yes | 445
  Dosing easy to take / convenient: No | 105
  Dosing easy to take / convenient: Missing | 2
  Effective to Treat Chest congestion:Very Satisfied | 108
  Effective to Treat Chest congestion:Somewhat Stfd | 386
  Effective to Treat Chest congestion:Somewhat Dstfd | 51
  Effective to Treat Chest congestion: Dissatisfied | 5
  Effective to Treat Chest congestion: Missing | 2
  Effective to Treat Chesty cough: Very Satisfied | 149
  Effective to Treat Chesty cough:Somewhat Satisfied | 361
  Effective to Treat Chesty cough: Somewhat Dstfd | 34
  Effective to Treat Chesty cough: Dissatisfied | 6
  Effective to Treat Chesty cough: Missing | 2
  Recommend to Family and friends: Yes | 305
  Recommend to Family and friends: Maybe | 216
  Recommend to Family and friends: No | 10
  Recommend to Family and friends: Missing | 21
  Mucinex as first choice | 171
  Mucinex as top two options | 133
  Mucinex as alternative, But not primary | 1

5. Secondary Outcome: Overall Assessment of the Study Medication by End of Study Investigator Questionnaire
Description: End of Study Investigator Questionnaire is a questionnaire provided at the end of study visit to the investigator (or sub-investigator as applicable) for overall assessment of the study medication across all patients treated by them.
  End of study investigator questionnaire was collected from 9 investigators.
  Mostly Satisfied(MS) Satisfied(Stfd) Very Satisfied(VS) Chest Congestion(CC) Chesty Cough(CCO) Difference(Diff) Between(b/w) Somewhat Agree(SA) Strongly Agree(StA) Upper respiratory tract infection(URTI) Optimal dosage(Opt dos) Cough preparations Available(CPA)
Time Frame: Up to Day 9
Population: Safety Population: All patients enrolled in the study were included for safety analyses.
Measure: Number; unit: Number of investigator
Arm/Group | Mucinex™
Number analyzed (Participants) | 552
Number of investigator
  Treatment outcome with URTIs taking Mucinex: MS | 2
  Treatment outcome with URTIs taking Mucinex: Stfd | 5
  Treatment outcome with URTIs taking Mucinex: VS | 2
  Patient satisfaction with the treatment of CC: NS | 1
  Patient satisfaction with the treatment of CC:Stfd | 5
  Patient satisfaction with the treatment of CC: VS | 3
  Patient satisfaction with the treatment of CCO: MS | 1
  Patient satisfaction with treatment of CCO:Stfd | 5
  Patient satisfaction with the treatment of CCO: VS | 3
  Reported Improvements: At 2 Days Of Treatment | 5
  Reported Improvements:Within 3 Days of Treatment | 4
  Treatment Diff b/w CC & CCO congestion: CC first | 7
  Treatment Diff b/w CC & CCO congestion:Cough first | 2
  Treatment recommend for CC with URTI Patient:Agree | 5
  Treatment recommend for CC with URTI Patient: SA | 1
  Treatment recommend for CC with URTI Patient: StA | 3
  Opt dos for treating CC compare to other CPA: No | 1
  Opt dos for treating CC compare to other CPA: Yes | 8

ADVERSE EVENTS:
Time Frame: Up to End of Study (Day 9)
Arm/Group | Mucinex™
All-Cause Mortality (participants affected / at risk) | 0/552
Serious Adverse Events (participants affected / at risk) | 0/552
Other Adverse Events (participants affected / at risk) | 28/552
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mucinex™ (N=552)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No